CLINICAL TRIAL: NCT06318260
Title: Haemodynamic Effects of Dobutamine in Patients With Wild-type Transthyretin Amyloid Cardiomyopathy (ATTRwt)
Acronym: DobATTR
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Steen Hvitfeldt Poulsen (Other)
Responsible Party: Sponsor-Investigator, Steen Hvitfeldt Poulsen, Professor, DMSc., Aarhus University Hospital Skejby
Organization: Aarhus University Hospital Skejby (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2023-508298-10-00
Record Dates: First submitted 2024-03-12; First posted 2024-03-19 (Actual); Last update posted 2024-04-17 (Actual); Status verified 2024-04

CONDITIONS: ATTR Amyloidosis Wild Type
Keywords: Cardiac amyloidosis; Inotropic; ATTR-CM; Transthyretin amyloid cardiomyopathy; Dobutamine; wild type ATTR
MeSH Terms: conditions — Amyloid Neuropathies, Familial | interventions — Dobutamine

STUDY DESIGN:
Intervention Model Description: Prospective, single-centre, one arm clinical explorative study, with consecutive enrolment.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- ATTRwt (Experimental): Dobutamine (Dobutrex®) infusion.
  Interventions: Drug: Dobutrex

INTERVENTIONS:
Drug: Dobutrex — Dobutamine (Dobutrex®) infusion. will be performed with a stepwise dobutamine dosage increase every 5 minutes (2,3,5,10,20 ug/kg/min). Dobutamine dosage will only be increased to 40 ug/kg/min in participants with ongoing beta-blocker treatment to ensure an appropriate dobutamine response. As dobutamine and its metabolites are excreted renally, the dose will be reduced to max 10 ug/kg/min in participants with eGFR below 30 mL/min/1,73 m2. Echocardiography, blood pressure, heart rate, and invasive pressure and flow measurements will be obtained before the infusion starts, at each infusion stage, and during the recovery period after the infusion is stopped.
  Other Names: Dobutamine

SUMMARY:
The goal of this clinical trial is to test the effects of the inotropic drug named dobutamine, in patients with wild-type Transthyretin Amyoid Cardiomyopathy (ATTRwt). The main questions it aims to answer are:

* What are the effects of increasing dosages of dobutamine infusion on cardiac output and filling pressures in patients with symptomatic ATTRwt.
* Safety of dobutamine infusion in this patient population.

Participants will be given increasing dosages of dobutamine infusion, and its effect on cardiac output and filling pressures will be assessed non-invasively by echocardiography, and invasively by right heart catheterization, simultaneously.

DETAILED DESCRIPTION:
AIMS

* To investigate the hemodynamic effects of increasing dosages of dobutamine infusion on cardiac output and filling pressures in patients with symptomatic ATTRwt, assessed simultaneously by right heart catheterization (RHC) and echocardiography.
* To assess the safety of dobutamine infusion in ATTRwt patients.

HYPOTHESIS

* Dobutamine infusion can increase myocardial contractility in patients with symptomatic ATTRwt with an increase of CO by 10%.
* The left ventricular filling pressure as expressed by the pulmonary artery wedge pressure (PAWP) and/or mean pulmonary artery pressure (mPAP) will decrease by ≥ 10% during increasing dobutamine dosages.
* Dobutamine is well-tolerated and safe to use in symptomatic ATTRwt patients.

MATERIALS AND METHODS

Study population Symptomatic participants with ATTRwt, age ≥ 65 years, who have reduced left ventricular ejection fraction (LVEF) and/or stroke volume index (SVI), without significant valvular diseases or severe coronary artery diseases.

Study design

Eligible patients will be assessed in the trial day (one day) as following:

Step1; Baseline assessment: Blood pressure, pulse and ECG will be obtained. All participants will also undergo a comprehensive resting transthoracic echocardiographic assessment according to current guidelines.

Step 2; Invasive right heart catheterization (RHC): The subjects will be instructed not to eat for 6 hours and not to drink for 2 hours before the procedure. RHC will be performed in the cardiac invasive laboratory using right internal jugular vein access. Rarely, right femoral vein access will be used, if the right internal jugular vein is difficult to canulate, as a result of anatomical anomalies or local skin or muscle deformities. A 7 Fr sheath will be inserted in the vein aseptic, and ultrasound guided in local anaesthesia. Subsequently, a pulmonary catheter (Swan-Ganz) will be advanced through the sheath guided by pressure waves and fluoroscopy, through the right atrium, the right ventricle, and ultimately in a stable position in the pulmonary artery (PA). The standard Swan-Ganz catheter is equipped with an inflatable balloon at the tip, which facilitates its placement into the PA through the flow of blood. The balloon, when inflated, causes the catheter to "wedge" in a small pulmonary blood vessel. While wedged, the catheter can provide an indirect measurement of the mean left atrium pressure. Central oxygenation of the blood (SvO2) and N-terminal pro-B-type natriuretic peptide (NT-proBNP) will be assessed from blood taken from the pulmonary artery at rest and at peak dobutamine infusion according to the protocol.

The PA catheter location will be confirmed with fluoroscopy before leaving the laboratory and both the sheath and the catheter will be fixed to the skin.

RHC is performed using a standard 7 Fr triple lumen Swan-Ganz catheter (Edwards Lifesciences, Irvine, California, USA).

The following parameters will be measured by RHC:

* PAWP
* Mean right atrial pressure
* Systolic and diastolic PA pressure
* mPAP
* CO All pressures at rest are measured at end-expiration as the average of five measurements. CO is measured using thermodilution methods as the average of at least four measurements not differing more than 10% and indexed to body surface area as the Cardiac Index (CI). SV is calculated as CO divided by heart rate.

Step 3; Dobutamine challenge:

Step 4; Recovery period: The pulmonary catheter and sheath will be removed after a-5-minute recovery period, right after obtaining the final images and invasive measurements. The participants will be observed for 2 hours after the end of the test and will be discharged if no complications arise. Blood sample will be taken to measure NT-proBNP after 1-2 hours after the end of dobutamine challenge.

The investigators expect the study will last for about 6-7 hours, including preparations, waiting time, the procedures themselves and the observation period.

ELIGIBILITY:
Inclusion Criteria:

1. ATTRwt, diagnosis confirmed by genetic testing, 99mTc-3,3-diphosphono-1,2-propanodicarboxylic acid (DPD) scintigraphy and/or endomyocardial biopsy.
2. Treated with loop diuretics.
3. New York Heart Association class II-IV.
4. Age ≥ 65 years.
5. Left ventricular ejection fraction (LVEF) < 50 % and/or SVI assessed by echocardiography < 35 ml/m2.
6. Thorough oral and written informed consent to participate in the study.

Exclusion Criteria:

1. Moderate to severe aortic stenosis (participants with aortic sclerosis will not be excluded).
2. Other significant valvular diseases.
3. Known severe coronary artery diseases: left main stem stenosis or 3-vessel disease, or recent acute myocardial infarction (< 4 weeks).
4. Contraindications to the use of dobutamine: Known allergy to dobutamine or sulfite, phaeochromocytoma or ventricular tachycardia (VT).
5. End stage renal disease (eGFR of less than 15 mL/min/1,73 m2).

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 35 (Estimated)
Dates: Start 2024-04-08 (Actual); Primary Completion 2025-09 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Cardiac output | Evaluated at every dobutamine dose-level, and at the end of infusion.
  Mean cardiac output increase by 10%, evaluated by the thermodynamic invasive methods.

SECONDARY OUTCOMES:
Increase in invasively measured SVI by ≥ 20%. | Evaluated at every dobutamine dose-level, and at the end of infusion.
Reduction in mean PAWP and/or mPAP by 10 %. | Evaluated at every dobutamine dose-level, and at the end of infusion.
Increase in LVEF and LV-global longitudinal strain (LV-GLS) of absolute 10 %. | Evaluated at every dobutamine dose-level, and at the end of infusion.
Correlation between echo- and invasive measured SVI, and CO. | Evaluated at every dobutamine dose-level, and at the end of infusion.
Rate of complications (i.e. Systolic blood pressure drop < 90 mmHg, arrhythmias)/symptomatic side effects. | Evaluated at every dobutamine dose-level, at the end of infusion, and during the 2 hours recovery period.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Cardiology, Aarhus University Hospital, Aarhus, Denmark